CLINICAL TRIAL: NCT03179020
Title: Cluster Randomized Trial Evaluating the Implementation of a Evidence Based Checklist for the Management of Potential Organ Donors
Brief Title: Donation Network to Optimize Organ Recovery Study
Acronym: DONORS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Moinhos de Vento (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DONORS Study
Record Dates: First submitted 2017-03-23; First posted 2017-06-07 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Brain Death; Organ Donation
Keywords: Intensive Care Units; Brain Death; Organ Donation; Family interview
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Intervention Model Description: In the present study ICUs will be randomized to manage potential organ donors through the use of a evidence-based checklist or to manage potential organ donors according usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Checklist ICUs (Experimental): Management of the potential donor guided by the use of an evidence-based checklist. This checklist is based on main recommendations of the Brazilian guideline for the management of potential multiple organ donors.
  Interventions: Other: Checklist use
- Usual Care ICUs (Active Comparator): Management of the potential donor according usual care.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Checklist use — Management of the potential donor guided by the use of an evidence-based checklist. This checklist is based on main recommendations of the Brazilian guideline for the management of potential multiple organ donors.
  Arms: Checklist ICUs
Other: Usual care — Management of the potential donor according usual care.
  Arms: Usual Care ICUs

SUMMARY:
This study consists in an cluster-randomized clinical trial involving near 60 Brazilian intensive care units (ICUs) with a high notification rate of potential donors of organs and tissues. ICUs will be randomized in a 1:1 ratio to manage potential organ donors through the use of a evidence-based checklist or to manage potential organ donors according usual care. The primary outcome is the rate of losses of potential donors due to cardiac arrest. Secondary outcome measures include number of effective organ donors and number of organs recovery per effective donor. The first subject was enrolled on June 20, 2018.

ELIGIBILITY:
Inclusion Criteria:

For ICUs:

* Adults ICUs reporting at least 10 potential valid donors (without clinical contraindications for donation) per year

For potential donor:

* Age of 14 years or older
* Suspected brain death after the first clinical test

Exclusion Criteria:

For ICUs:

* Coronary units, intermediate units, emergency services
* ICUs that use checklist for the management of the potential donors

For potential donors:

* Age >90 years
* HIV
* Metastatic cancer
* Uncontrolled sepsis
* Acute hepatitis
* Malaria
* Acute viral infections
* Cryptococcal meningoencephalitis and prion diseases
* Active tuberculosis treated less than 2 months
* Colonization of the donor by bacteria without any option of antibiotic treatment
* History of breast tumor, melanoma, soft tissue sarcoma or hematologic neoplasia, WHO Group 3 primary tumors

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1535 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Losses of potential donors due to cardiac arrest | This event will be evaluated from the date of study subject enrollment until the date of organ recovery or end of brain death protocol (for cases of family refusal or contraindications to organ recovery) assessed up to 14 days
  Proportion of losses of potential donors due to cardiac arrest

SECONDARY OUTCOMES:
Effective organ donor | This event will be evaluated from the date of study subject enrollment until the date of organ recovery or end of brain death protocol (for cases of family refusal or contraindications to organ recovery) assessed up to 14 days
  Proportion of Effective organ donors
Organ recovery per effective donor | This event will be evaluated from the date of study subject enrollment until the date of organ recovery assessed up to 14 days
  Number of organs recovery per effective donor

CONTACTS AND LOCATIONS:
Overall Officials: Glauco Westphal, MD, PhD, Principal Investigator — Hospital Moinhos de Vento; Regis G Rosa, MD, PhD, Study Director — Hospital Moinhos de Vento
Locations (63):
- Brazil (63):
  - Hospital das Clínicas de Rio Branco, Rio Branco, Acre
  - Hospital de Urgência e Emergência de Rio Branco, Rio Branco, Acre
  - Hospital Geral Prof. Osvaldo Brandão Vilela, Maceió, Alagoas
  - Hospital de Pronto Socorro Dr. João Lúcio Pereira Machado, Manaus, Amazonas
  - Hospital Geral de Fortaleza, Fortaleza, Ceará
  - Hospital Insituto Dr José Frota, Fortaleza, Ceará
  - Hospital Regional do Cariri, Juazeiro do Norte, Ceará
  - Hospital Regional Tarcisio de Vasconcelos Maia, Mossoró, Ceará
  - Hospital Regional Norte, Sobral, Ceará
  - Santa Casa de Misericórdia de Sobral, Sobral, Ceará
  - Hospital Estadual de Urgência e Emergência de Vitória, Vitória, Espírito Santo
  - Hospital Geral Cleriston Andrade, Feira de Santana, Estado de Bahia
  - Hospital de Base do Distrito Federal, Brasília, Federal District
  - Hospital de Urgência de Goiânia, Goiânia, Goiás
  - Hospital Dr Carlos Macieira, São Luís, Maranhão
  - Socorrão I - Hospital Municipal Djalma Marques, São Luís, Maranhão
  - Santa Casa de Campo Grande, Campo Grande, Mato Grosso do Sul
  - Hospital das Clinicas das Minas Gerais, Belo Horizonte, Minas Gerais
  - Hospital João XXIII Fundação Hospitalar do Estado de Minas Gerais, Belo Horizonte, Minas Gerais
  - Hospital Universitário Ciências Médicas, Belo Horizonte, Minas Gerais
  - Santa Casa de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Hospital Norte Paranaense, Arapongas, Paraná
  - Hospital e Maternidade Angelina Caron, Campina Grande do Sul, Paraná
  - Hospital Nossa Senhora do Rocio de Campo Largo, Campo Largo, Paraná
  - Hospital Universitário de Cascavel do Oeste do Paraná, Cascavel, Paraná
  - Hospital Municipal Padre Germano Lauk, Foz do Iguaçu, Paraná
  - Hospital São Vicente de Paulo Guarapuava, Guarapuava, Paraná
  - Hospital Evangélico de Londrina, Londrina, Paraná
  - Hospital Universitário Regional do Norte do Paraná, Londrina, Paraná
  - Hospital Santa Rita de Maringá, Maringá, Paraná
  - Hospital Universitário de Maringá, Maringá, Paraná
  - Irmandade Santa Casa de Misericórdia de Maringá, Maringá, Paraná
  - Hospital Bom Jesus de Ponta Grossa, Ponta Grossa, Paraná
  - Hospital Universitario Regional dos Campos Gerais, Ponta Grossa, Paraná
  - Hospital Bom Jesus de Toledo, Toledo, Paraná
  - Alberto Urquiza Wanderley - Unimed João Pessoa, João Pessoa, Paraíba
  - Hospital de Ensino Doutor Washington Antônio de barros, Petrolina, Pernambuco
  - Hospital da Restauração, Recife, Pernambuco
  - Hospital Geral de Nova Iguaçu, Nova Iguaçu, Rio de Janeiro
  - Hospital de Canoas, Canoas, Rio Grande do Sul
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital Universitário São Francisco de Paula, Pelotas, Rio Grande do Sul
  - Hospital Cristo Redentor, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Pronto Socorro de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Irmandade da Santa Casa de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Pronto Socorro João Paulo II, Porto Velho, Rondônia
  - Hospital de Urgência de Sergipe, Aracaju, Sergipe
  - Hospital das Clínicas de Botucatu, Botucatu, São Paulo
  - Hospital Universitário São Francisco da Providência de Deus de Bragança Paulista, Bragança Paulista, São Paulo
  - Hospital Municipal Irmã Dulce, Praia Grande, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto, São Paulo
  - Casa de Saúde de Santos, Santos, São Paulo
  - Hospital de Base de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Irmandade Santa Casa de Misericórdia de Sorocaba, Sorocaba, São Paulo
  - Hospital Regional do Vale do Paraíba, Taubaté, São Paulo
  - Hospital Estadual Getúlio Vargas, Rio de Janeiro
  - Hospital Beneficência Portuguesa de São Paulo, São Paulo
  - Hospital Geral de Taipas, São Paulo
  - Hospital Paulistano, São Paulo
  - Hospital São Paulo, São Paulo
  - Irmandade da Santa Casa de Misericórdia de São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Westphal GA, Robinson CC, Giordani NE, Teixeira C, Rohden AI, Dos Passos Gimenes B, Guterres CM, Madalena IC, Andrighetto LV, Souza da Silva S, Barbosa da Silva D, Sganzerla D, Cavalcanti AB, Franke CA, Bozza FA, Machado FR, de Andrade J, Pontes Azevedo LC, Schneider S, Orlando BR, Grion CMC, Bezerra FA, Roman FR, Leite FO Jr, Ferraz Siqueira IL, Oliveira JFP, de Oliveira LC Jr, de Melo MFRB, Leal PBGP, Diniz PC, Moraes RB, Salomao Pontes DF, Araujo Queiroz JE, Hammes LS, Meade MO, Rosa RG, Falavigna M; DONORS (Donation Network to Optimize Organ Recovery Study) Investigators and the BRICNet (Brazilian Research in Intensive Care Network). Evidence-Based Checklist to Delay Cardiac Arrest in Brain-Dead Potential Organ Donors: The DONORS Cluster Randomized Clinical Trial. JAMA Netw Open. 2023 Dec 1;6(12):e2346901. doi: 10.1001/jamanetworkopen.2023.46901. PMID 38095899
- [Derived] Giordani NE, Robinson CC, Westphal GA, Rosa RG, Sganzerla D, Cavalcanti AB, Machado FR, Azevedo LCP, Bozza FA, Teixeira C, de Andrade J, Franke CA, Guterres CM, Madalena IC, Rohden AI, da Silva SS, Andrighetto LV, Rech GS, Gimenes BDP, Hammes LS, Pontes DFS, Meade MO, Falavigna M. Statistical analysis plan for a cluster-randomised trial assessing the effectiveness of implementation of a bedside evidence-based checklist for clinical management of brain-dead potential organ donors in intensive care units: DONORS (Donation Network to Optimise Organ Recovery Study). Trials. 2020 Jun 17;21(1):540. doi: 10.1186/s13063-020-04457-1. PMID 32552839
- [Derived] Westphal GA, Robinson CC, Biasi A, Machado FR, Rosa RG, Teixeira C, de Andrade J, Franke CA, Azevedo LCP, Bozza F, Guterres CM, da Silva DB, Sganzerla D, do Prado DZ, Madalena IC, Rohden AI, da Silva SS, Giordani NE, Andrighetto LV, Benck PS, Roman FR, de Melo MFRB, Pereira TB, Grion CMC, Diniz PC, Oliveira JFP, Mecatti GC, Alves FAC, Moraes RB, Nobre V, Hammes LS, Meade MO, Nothen RR, Falavigna M; DONORS (Donation Network to Optimise Organ Recovery Study) Investigators and the BRICNet. DONORS (Donation Network to Optimise Organ Recovery Study): Study protocol to evaluate the implementation of an evidence-based checklist for brain-dead potential organ donor management in intensive care units, a cluster randomised trial. BMJ Open. 2019 Jun 25;9(6):e028570. doi: 10.1136/bmjopen-2018-028570. PMID 31243035